CLINICAL TRIAL: NCT01840982
Title: A Randomized, Crossover Clinical Trial, The Effects of Mixed Grain on Blood Glucose and Insulin in Healthy Male
Brief Title: The Effects of Mixed Grain on Blood Glucose and Insulin in Healthy Male
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Director, Chonbuk National University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CTCF2_2010_MC_2
Record Dates: First submitted 2013-04-05; First posted 2013-04-26 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Healthy People; Diabetes Mellitus, Type 2
Keywords: Mixed grains; Glycemic index; Giant embryonic brown rice; Giant embryonic rice; diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Giant embryonic brown rice (Experimental)
  Interventions: Dietary Supplement: Mixed grain 1
- Giant embryonic rice (Experimental)
  Interventions: Dietary Supplement: Mixed grain 2
- White rice (Active Comparator)
  Interventions: Dietary Supplement: White rice
- Glucose solution (Active Comparator)
  Interventions: Other: Glucose solution

INTERVENTIONS:
Dietary Supplement: Mixed grain 1 — All test foods contained 50 g available carbohydrate from the test food products. A glass of 200 ml water was served together with the clinical trial food, and the participants were instructed to ingest the breakfast with 15 min.
  Other Names: Mixed grain 1 (Giant embryonic brown rice) diet
  Arms: Giant embryonic brown rice
Dietary Supplement: Mixed grain 2 — All test foods contained 50 g available carbohydrate from the test food products. A glass of 200 ml water was served together with the clinical trial food, and the participants were instructed to ingest the breakfast with 15 min.
  Other Names: Mixed grain 2 (Giant embryonic rice) diet
  Arms: Giant embryonic rice
Dietary Supplement: White rice — All test foods contained 50 g available carbohydrate from the test food products. A glass of 200 ml water was served together with the clinical trial food, and the participants were instructed to ingest the breakfast with 15 min.
  Other Names: control diet
  Arms: White rice
Other: Glucose solution — All test foods contained 50 g available carbohydrate from the test food products.
  Other Names: Reference diet
  Arms: Glucose solution

SUMMARY:
This study was an open, 4-treatment, 5-sequence, 5-day cross-over randomized design clinical trial to evaluate the efficacy of mixed grain on blood glucose, insulin and Glycemic index(GI) in healthy males.

DETAILED DESCRIPTION:
After a 12-hour fast, oral glucose or meal tolerance test was performed with blood samples drawn at time 0, 15, 30, 45, 90, 120, 150, and 180 min.

1. Serum levels of glucose, insulin, and C-peptide were analyzed by biochemical autoanalyzer. The area under the curve (AUC) changes in blood glucose were computed by the trapezoidal method.
2. Glycemic index(GI): the area under the glucose response curve after consumption of a test food divided by the area under the curve after consumption of a control food containing the same amount of carbohydrate and calculated using 50 g glucose as the reference.

ELIGIBILITY:
Inclusion Criteria:

* Males, 19~60years old
* Bodyweight was more than 50 kg with ideal body weight within ±30%
* Less than 100 mg/dl in fasting blood glucose and less than 140 mg/dl in an oral glucose tolerance test (OGTT)
* Able to give informed consent

Exclusion Criteria:

* Major medical illness such as cardiovascular, neurologic, psychiatric, renal, pulmonary and hepatic diseases
* History of disease that could interfere with the test products or impede their absorption such as gastrointestinal disease or gastrointestinal surgery
* Medical or psychological conditions deemed by the investigators to interfere with successful participation in the study
* Poor vital sign (systolic blood pressure: below 100 mmHg or above 150 mmHg, diastolic blood pressure: below 65 mmHg or above95 mmHg)
* Allergic or hypersensitive to any of the ingredients in the test products; treated with any drug within past 2 weeks
* Participation in any other clinical trials within past 2 months
* Alcohol consumption above 21 units per week or abnormal screening laboratory test
* Being judged by the responsible physician of the local study center as unfit to participate in the study

Ages: 19 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2015-03-25 (Actual)

PRIMARY OUTCOMES:
1. Glycemic index(GI) 2. Glucose, insulin AUC(incremental area under the curve) 3. C-peptide | 2 hour postprandial blood glucose, insulin, c-peptide
  1. Glycemic index (GI) was defined as the area under the glucose response curve after consumption of a test food divided by the area under the curve after consumption of a control food containing the same amount of carbohydrate and calculated using 50 g glucose as the reference. Plasma glucose will be measured at baseline, 15, 30, 45, 60, 90, and 120 minutes post ingestion of each test solution.
     GI= (incremental blood glucose area of test meal/incremental area of glucose) × 100
  2. Plasma glucose and insulin will be measured at baseline, 15, 30, 45, 60, 90, 120, 180 and 240 minutes post ingestion of each test solution, and area under the curve will be calculated.
  3. Plasma c-peptide will be measured at baseline, 120 minutes post ingestion of each test solution.

SECONDARY OUTCOMES:
Homeostatic model assessment-insulin resistance(HOMA-IR), quantitative insulin sensitivity check index(QUICKI), Insulinogenic index(IGI) | fasting and postprandial (different times for 30min)
  1. HOMA-IR={fasting insulin(µU/㎖) x fasting glucose(m㏖/L)}/22.5
  2. QUICKI=1/log(insulin 0min)-log(glucose 0min)
  3. IGI=(insulin 30min-fasting insulin)/(glucose 30min-fasting glucose)

CONTACTS AND LOCATIONS:
Overall Officials: Soo-Wan Chae, MD., PhD, Study Director — Chonbuk National University Hospital
Locations (1):
- Clinical Trial Center for Functional Foods; Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea